CLINICAL TRIAL: NCT04097223
Title: Real-world Treatment of Newly Diagnosed COPD Patients: A Retrospective German Claims Data Analysis
Brief Title: A Study Based on Health Insurance Data About the Treatment of Patients Who Have Been Newly Diagnosed With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1237-0092
Record Dates: First submitted 2019-09-04; First posted 2019-09-20 (Actual); Results first posted 2021-09-09 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with Pulmonary Disease, Chronic Obstructive

SUMMARY:
A retrospective analysis study in COPD patients for an exact follow-up period of 12 months (in subgroup analyses: 24 and 36 months); censoring of patients will only be done in case a patient died during the respective follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* All patients who were continuously insured by the sickness fund for the entire period (01/01/2013-30/06/2018) or, in case a patient deceased after index date, for the time until death
* A patient will be included as an incident COPD patient if either a hospital documented at least one COPD diagnosis (International Statistical Classification of Diseases and Related Health Problems (ICD-10 J 44.-) or a specialist (pneumologist) documented at least 2 confirmed COPD diagnoses (above ICD-10) code) in two different quarters; the first of the above diagnoses is defined as index diagnosis; inclusion period is defined as lasting from 01/01/2014 until 30/06/2017
* Patients should not have received any COPD diagnosis (ICD-10 J44.-) or any COPD-associated medication in the 12 months pre-index period
* Patient should have, at date of incident COPD diagnosis (index date), an age of at least 40 years

Exclusion Criteria:

* Patients received , at least one confirmed inpatient asthma diagnosis or two confirmed outpatient diagnoses of asthma (ICD-10: J45) by pneumologists

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A retrospective analysis of patients with Chronic Obstructive Pulmonary Disease (COPD) based on current German COPD guidleines.
Sampling Method: Non-Probability Sample
Enrollment: 17464 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for pharmacoeconomics and pharmaceutical logistics e.V (IPAM), Wismar, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A retrospective, non-interventional, longitudinal study including real-world data from german claims data (2015-2018) to describe the real-world drug treatment in patients of newly diagnosed chronic obstructive pulmonary disease (COPD).
Pre-assignment Details: Only subjects that met all inclusion and none of the exclusion criteria were included in the study.
Groups:
- COPD-FULL Sample: Patients with incident chronic obstructive pulmonary disease (COPD) between April 2015 and March 2018 from German claims database were followed for up to 48 months. Patients were censored in case of death or loss to follow-up.
Period: Overall Study
Arm/Group | COPD-FULL Sample
Started | 17464
Completed | 17464
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with newly diagnosed chronic obstructive pulmonary disease (Incident COPD patients).
Arm/Group | COPD-FULL Sample
Number analyzed (Participants) | 17464
Age, Continuous [Mean (Standard Deviation); unit: Years] | 71.5 (12.3)
Sex/Gender, Customized [Number; unit: Percentage of participants]
  Female | 41.4
  Male | 58.6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Description of Real-life Drug Treatment After Incident Diagnosis - COPD-12 Sample
Description: Description of real-life drug treatment in patients with newly diagnosed (incident) chronic obstructive pulmonary disease (COPD) in the first 12 months after the index date (date of incident (first) diagnosis of COPD). Reported is the percentage of patients per treatment and therapy line. The arms are not mutually exclusive, as patients switched to another treatment during follow-up period.
  COPD-12 sample: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with follow-up of 12 months since index date (COPD-12).
  LABA: Long-acting beta agonist; LAMA: Long-acting muscarinic antagonist, ICS: Inhaled corticosteroids.
Time Frame: Up to 12 months after the index date.
Population: All patients included in the COPD-12 sample, who received any long term-COPD treatment. Patients are reported by therapy line (arms are not mutually exclusive). The number of patients who received COPD-12 Fourth Line Therapy is less than 5% of the patient population (N=8238). As defined in the protocol, data collected only for treatment pattern combinations that were observed in >5% in patient population.
Measure: Number; unit: Percentage of Patients
Groups:
- COPD-12 - First Line Therapy: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with follow-up of 12 months since index date, who received first line therapy.
- COPD-12 - Second Line Therapy: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with follow-up of 12 months since index date, who received second line therapy.
- COPD-12 - Third Line Therapy: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with follow-up of 12 months since index date, who received third line therapy.
- COPD-12 - Fourth Line Therapy: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with follow-up of 12 months since index date, who received fourth line therapy.
Arm/Group | COPD-12 - First Line Therapy | COPD-12 - Second Line Therapy | COPD-12 - Third Line Therapy | COPD-12 - Fourth Line Therapy
Number analyzed (Participants) | 8238 | 1325 | 213 | 0
Percentage of Patients
  LABA + LAMA | 35.6 | 30.3 | 29.1 |
  LAMA | 25.0 | 11.3 | 10.3 |
  LAMA + ICS | 16.3 | 14.3 | 13.6 |
  LABA | 8.5 | 5.4 | 5.6 |
  LABA + LAMA + ICS | 8.1 | 24.8 | 25.8 |
  ICS | 4.2 | 4.8 | 6.1 |
  Other (Methylxanthine, LAMA+ICS, LABA+LAMA+Methyl-xanthine) | 2.3 | 9.0 | 9.4 |

2. Primary Outcome: Description of Real-life Drug Treatment After Incident Diagnosis - COPD-24 Sample
Description: Description of real-life drug treatment in patients with newly diagnosed (incident) chronic obstructive pulmonary disease (COPD) in the first 24 months after the index date (date of incident (first) diagnosis of COPD). Reported is the percentage of patients per treatment and therapy line. The arms are not mutually exclusive, as patients switched to another treatment during follow-up period.
  COPD-24 sample: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with follow-up of 24 months since index date (COPD-24).
  LABA: Long-acting beta agonist; LAMA: Long-acting muscarinic antagonist, ICS: Inhaled corticosteroids.
Time Frame: Up to 24 months after the index date.
Population: All patients included in the COPD-24 sample, who received any long term-COPD treatment. Patients are reported by therapy line (arms are not mutually exclusive).
Measure: Number; unit: Percentage of Patients
Groups:
- COPD-24 - First Line Therapy: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with follow-up of 24 months since index date, who received first line therapy.
- COPD-24 - Second Line Therapy: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with follow-up of 24 months since index date, who received second line therapy.
- COPD-24 - Third Line Therapy: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with follow-up of 24 months since index date, who received third line therapy.
- COPD-24 - Fourth Line Therapy: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with follow-up of 24 months since index date (COPD-24), who received fourth line therapy.
Arm/Group | COPD-24 - First Line Therapy | COPD-24 - Second Line Therapy | COPD-24 - Third Line Therapy | COPD-24 - Fourth Line Therapy
Number analyzed (Participants) | 5484 | 1411 | 432 | 126
Percentage of Patients
  LABA + LAMA | 34.4 | 30.6 | 25.0 | 25.4
  LAMA | 24.6 | 11.6 | 11.3 | 10.3
  LAMA + ICS | 17.3 | 15.2 | 13.7 | 15.1
  LABA | 9.2 | 5.0 | 5.6 | 4.8
  LABA + LAMA + ICS | 7.5 | 24.9 | 28.7 | 23.9
  ICS | 4.9 | 4.6 | 4.9 | 4.8
  Other (Methylxanthine, LAMA+ICS, LABA+LAMA+Methyl-xanthine) | 2.2 | 8.2 | 10.9 | 15.9

3. Primary Outcome: Description of Real-life Drug Treatment After Incident Diagnosis - COPD-36 Sample
Description: Description of real-life drug treatment in patients with newly diagnosed (incident) chronic obstructive pulmonary disease (COPD) in the first 36 months after the index date (date of incident (first) diagnosis of COPD). Reported is the percentage of patients per treatment and therapy line. The arms are not mutually exclusive, as patients switched to another treatment during follow-up period.
  COPD-36 sample: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with follow-up of 36 months since index date (COPD-36).
  LABA: Long-acting beta agonist; LAMA: Long-acting muscarinic antagonist, ICS: Inhaled corticosteroids.
Time Frame: Up to 36 months after the index date.
Population: All patients included in the COPD-36 sample, who received any long term-COPD treatment. Patients are reported by therapy line (arms are not mutually exclusive).
Measure: Number; unit: Percentage of Patients
Groups:
- COPD-36 - First Line Therapy: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with follow-up of 36 months since index date, who received first line therapy.
- COPD-36 - Second Line Therapy: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with follow-up of 36 months since index date, who received second line therapy.
- COPD-36 - Third Line Therapy: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with follow-up of 36 months since index date, who received third line therapy.
- COPD-36 - Fourth Line Therapy: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with follow-up of 36 months since index date, who received fourth line therapy.
Arm/Group | COPD-36 - First Line Therapy | COPD-36 - Second Line Therapy | COPD-36 - Third Line Therapy | COPD-36 - Fourth Line Therapy
Number analyzed (Participants) | 2445 | 801 | 300 | 119
Percentage of Patients
  LABA + LAMA | 31.3 | 32.2 | 27.7 | 29.4
  LAMA | 25.2 | 12.5 | 12.3 | 4.2
  LAMA + ICS | 17.8 | 15.5 | 13.3 | 16.0
  LABA | 9.3 | 6.1 | 7.0 | 5.0
  LABA + LAMA + ICS | 7.9 | 20.6 | 24.3 | 21.0
  ICS | 6.3 | 4.9 | 5.0 | 5.0
  Other (Methylxanthine, LAMA+ICS, LABA+LAMA+Methyl-xanthine) | 2.2 | 8.2 | 10.3 | 19.3

4. Primary Outcome: Number of Observed Treatment Lines - COPD-12, COPD-24, COPD-36 and COPD-FULL Sample
Description: Number of treatment lines an observed patient received in the first 12/24/36 and 48 months after incident diagnosis.
Time Frame: Up to 12, 24, 36 and 48 months after index date for COPD-12, COPD-24, COPD-36 and COPD-FULL sample respectively.
Population: All patients with newly diagnosed (incident) COPD and who received any long-term COPD treatment. Incident COPD-patients are reported by follow-up period (12, 24, 36 and 48 months). Arms are not mutually exclusive.
Measure: Mean (Standard Deviation); unit: Treatment lines
Groups:
- COPD-12 Sample: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with a follow-up of 12 months since index date (COPD-12).
- COPD-24 Sample: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with a follow-up of 24 months since index date (COPD-24).
- COPD-36 Sample: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with a follow-up of 36 months since index date (COPD-36).
Arm/Group | COPD-FULL Sample | COPD-12 Sample | COPD-24 Sample | COPD-36 Sample
Number analyzed (Participants) | 9981 | 8238 | 5484 | 2445
Treatment lines | 1.39 (0.83) | 1.43 (0.86) | 1.51 (0.97) | 1.61 (1.06)

5. Primary Outcome: Percentage of Patients Per Most Frequently Prescribed Non-COPD Agents in COPD-FULL, COPD-12, COPD-24 and COPD-36 Samples
Description: Percentage of participants per most frequently prescribed non-COPD agents in the first 12/24/36 and 48 months after incident diagnosis.
  GERD: Gastroesophageal reflux disease.
Time Frame: Up to 12, 24, 36 and 48 months after index date for COPD-12, COPD-24, COPD-36 and COPD-FULL sample respectively.
Population: All patients with newly diagnosed (incident) chronic obstructive pulmonary disease. Incident COPD-patients were reported by follow-up time (12, 24, 36 and 48 months). Arms are not mutually exclusive.
Measure: Number; unit: Percentage of participants
Arm/Group | COPD-FULL Sample | COPD-12 Sample | COPD-24 Sample | COPD-36 Sample
Number analyzed (Participants) | 17464 | 14213 | 8804 | 3804
Percentage of participants
  Beta-blocking agents | 45.9 | 51.9 | 55.6 | 57.8
  Anti-thrombotic agents | 41.1 | 45.0 | 49.4 | 52.6
  High-ceiling diurectis | 37.9 | 40.4 | 43.3 | 43.7
  Drugs for peptic ulcer or GERD | 37.9 | 41.8 | 48.0 | 53.2
  Other analgesics & antipyretics | 20.3 | 20.5 | 29.7 | 36.7

6. Secondary Outcome: Percentage of Incident COPD-patients With Initial Treatment Not in Line Treatment Guideline - COPD-12 Sample
Description: Percentage of incident chronic obstructive pulmonary disease (COPD) patients with initial drug treatment not in line with 2012/2018 german guidelines. Results are reported for COPD-12 sample. According to guidelines the initial treatment with long-acting bronchodilators should generally not include use of Inhaled corticosteroids (ICS) (both guidelines). Based on the 2012 guideline, a therapy with long-acting bronchodilators should not start with a combination of Long-acting beta agonist (LABA) + Long-acting muscarinic antagonist (LAMA) or triple therapy of LAMA+LABA+ ICS.
Time Frame: At index date.
Population: All patients with newly diagnosed chronic obstructive pulmonary disease (COPD), with a follow-up of 12 months since index date (COPD-12).
Measure: Number; unit: Percentage of Patients
Arm/Group | COPD-12 Sample
Number analyzed (Participants) | 14213
Percentage of Patients
  Any ICS containing therapy | 14.1
  LAMA + LABA combination | 22.7
  LABA + LAMA + ICS | 4.7

7. Secondary Outcome: Percentage of Incident COPD-patients With Treatment Not in Line Treatment Guideline - COPD-12 Sample (Triple Therapy)
Description: Percentage of incident chronic obstructive pulmonary disease (COPD) patients with drug treatment not in line with 2012/2018 german guidelines. Results are reported for COPD-12 sample, who received triple therapy (Long-acting beta agonist (LABA) + Long-acting muscarinic antagonist (LAMA) + Inhaled corticosteroids (ICS)) within the first 12 months after incident diagnosis.
  According to both guidelines (2012/2018) a triple combination treatment should not be prescribed if only 1 or less confirmed outpatient diagnoses and no inpatient diagnosis of a COPD exacerbation (ICD-10 J44.1) before date of prescription of a triple therapy.
  FEV1: Forced expiratory volume (in 1 second).
Time Frame: At first day of triple therapy prescription, (which is not the index date), up to 12 months.
Population: All patients included in the COPD-12 sample, who received triple therapy within the first 12 months after incident COPD.
Measure: Number; unit: Percentage of Patients
Arm/Group | COPD-12 Sample
Number analyzed (Participants) | 1019
Percentage of Patients
  ≤1 Outpatient diagnosis and no inpatient diagnosis indicating COPD related exacerbation | 69
  Documented FEV1 ≥50% value | 75

8. Secondary Outcome: Percentage of Incident COPD-patients With Treatment Not in Line Treatment Guideline - COPD-12 Sample (Escalation Therapy)
Description: Percentage of incident chronic obstructive pulmonary disease (COPD) patients with drug treatment not in line with 2012/2018 german guidelines. Results are reported for patients in COPD-12 sample, with treatment escalation (mono therapy to Long-acting beta agonist (LABA)/ Long-acting muscarinic antagonist (LAMA)/ Inhaled corticosteroids (ICS), LABA/ICS or LAMA/LABA to LABA/LAMA/ICS) within the first 12 months after index date.
  According to guidelines patients should not receive a treatment intensification without any previous visit of a pneumologist or hospital (same quarter or previous quarter).
Time Frame: Up to 12 months after index date.
Population: All patients in the COPD-12 sample with treatment escalation in the first 12 months after index date.
Measure: Number; unit: Percentage of Patients
Arm/Group | COPD-12 Sample
Number analyzed (Participants) | 513
Percentage of Patients | 13

9. Secondary Outcome: Percentage of Patients With Exacerbations After Incident Diagnosis in COPD-12, COPD-24, COPD-36 and COPD-FULL Samples
Description: Description of exacerbation (severe exacerbations associated with hospitalizations) frequency of patients with newly diagnosed (incident) chronic obstructive pulmonary disease (COPD) in the first 12, 24, 36 and 48 months after incident diagnosis.
  Reported is the percentage of patients with exacerbations by the following categories:
  More or equal than one exacerbation (≥ 1) ;
  1. exacerbation;
  2. exacerbations;
  3. exacerbations; more than 3 exacerbations (> 3 exacerbations).
Time Frame: Up to 12,24, 36 and 48 months after index date, for COPD-12, COPD-24, COPD-36 and COPD-FULL sample respectively.
Population: All patients with newly diagnosed (incident) chronic obstructive pulmonary disease. Incident COPD-patients were reported by follow-up time (12, 24, 36 and 48 months), arms are not mutually exclusive.
Measure: Number; unit: Percentage of participants
Groups:
- Overall COPD-sample: All observed patients with incident chronic obstructive pulmonary disease (COPD) between April 2015 and March 2018 from German claims database. Patients were censored in case of death or loss to follow-up.
Arm/Group | Overall COPD-sample | COPD-12 Sample | COPD-24 Sample | COPD-36 Sample
Number analyzed (Participants) | 17464 | 14213 | 8804 | 3804
Percentage of participants
  ≥ 1 exacerbation | 12.0 | 10.1 | 11.0 | 12.2
  1 exacerbation | 9.8 | 8.0 | 8.5 | 9.5
  2 exacerbation | 1.5 | 1.4 | 1.7 | 1.8
  3 exacerabation | 0.4 | 0.4 | 0.4 | 0.5
  ≥ 3 exacerbation | 0.3 | 0.3 | 0.4 | 0.4

10. Secondary Outcome: Number of Yearly Visits Per Outpatient Treatment in COPD-12, COPD-24 and COPD-36 Samples
Description: Description of health-care resource use (HCRU) in the first 12/24/36 months after incident diagnosis - Number of yearly visits (outpatient treatment).
  Following categories are reported:
  Number of yearly general practitioner (GP) visits; Number of yearly pulmonologist visits; Number of yearly other specialist (primarily Ophthalmologist, Ear, Nose and Throat (ENT) specialist and Orthopedist) visits.
  Reported is the average number of yearly visits, per observed patient year.
Time Frame: Up to 12, 24 and 36 months after index date for COPD-12, COPD-24 and COPD-36 sample respectively.
Population: Patients with newly diagnosed (incident) chronic obstructive pulmonary disease (COPD). Incident COPD-patients were reported by follow-up time (COPD-12, COPD-24, COPD-36) and available Disease Management Program (DMP) data. Arms are not mutually exclusive.
Measure: Mean (Standard Deviation); unit: Yearly visits
Groups:
- COPD-12 Sample With DMP Data: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with a follow-up of 12 months since index date and with available Data Management Program (DMP) data (at least one entry during 3 months after index date). (COPD DMP-12).
Arm/Group | COPD-12 Sample | COPD-24 Sample | COPD-36 Sample | COPD-12 Sample With DMP Data
Number analyzed (Participants) | 14213 | 8804 | 3804 | 1434
Yearly visits
  Number of yearly GP visits | 4.58 (1.91) | 4.48 (1.69) | 4.45 (1.61) | 4.30 (1.91)
  Number of yearly pulmonologist visits | 1.08 (1.57) | 1.00 (1.37) | 0.92 (1.27) | 2.76 (1.57)
  Number of yearly other specialist visits | 7.73 (5.84) | 7.66 (5.50) | 7.67 (5.35) | 8.11 (5.84)

11. Secondary Outcome: Number of Yearly Hospitalizations in COPD-12, COPD-24 and COPD-36 Samples
Description: Description of health-care resource use in the first 12/24/36 months after incident diagnosis: Number of yearly hospitalizations (inpatient treatment).
  Following categories of inpatient treatment are reported:
  Number of yearly hospitalizations with exacerbations (J44.1); Number of yearly hospitalizations with exacerbations, any COPD diagnosis (J44); Number of yearly hospitalizations with non-COPD diagnosis. Results are reported by follow-up time and available Disease Management Program (DMP) data.
Time Frame: Up to 12, 24 and 36 months after index date for COPD-12, COPD-24 and COPD-36 sample respectively.
Population: Patients with newly diagnosed (incident) chronic obstructive pulmonary disease (COPD). Incident COPD-patients were reported by follow-up time (12, 24 and 36 months) and available Disease Management Program (DMP) data. Arms are not mutually exclusive.
Measure: Mean (Standard Deviation); unit: Yearly hospitalizations
Groups:
- COPD-12 Sample With DMP Data: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with a follow-up of 12 months since index date and with available Data Monitoring Program (DMP) data (at least one entry during 3 months after index date). (COPD DMP-12).
- COPD-24 Sample With DMP Data: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with a follow-up of 24 months since index date and with available Data Monitoring Program (DMP) data (at least one entry during 3 months after index date). (COPD DMP-24).
- COPD-36 Sample With DMP Data: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with a follow-up of 36 months since index date and with available Data Monitoring Program (DMP) data (at least one entry during 3 months after index date). (COPD DMP-36).
Arm/Group | COPD-12 Sample | COPD-24 Sample | COPD-36 Sample | COPD-12 Sample With DMP Data | COPD-24 Sample With DMP Data | COPD-36 Sample With DMP Data
Number analyzed (Participants) | 14213 | 8804 | 3804 | 1434 | 973 | 445
Yearly hospitalizations
  Yearly hospitalizations with exacerbation (J44.1) | 0.09 (0.34) | 0.06 (0.22) | 0.04 (0.16) | 0.11 (0.35) | 0.07 (0.24) | 0.05 (0.15)
  Yearly hospitalizations - any COPD diagnosis (J44) | 0.17 (0.45) | 0.10 (0.28) | 0.08 (0.21) | 0.18 (0.44) | 0.12 (0.30) | 0.09 (0.21)
  Yearly hospitalizatons with non-COPD diagnosis | 2.02 (2.08) | 1.38 (1.46) | 1.17 (1.22) | 1.09 (1.54) | 0.84 (1.06) | 0.74 (0.95)

12. Secondary Outcome: Time to First All-cause Hospitalization in COPD-12, COPD-24, COPD-36 Samples
Description: Description of health-care resource use in the first 12/24/36 months after incident diagnosis in patients with chronic obstructive pulmonary disease (COPD). Reported is time to first all-cause hospitalization in days (inpatient treatment).
Time Frame: Up to 12, 24 and 36 months after index date for COPD-12, COPD-24 and COPD-36 sample respectively.
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: Days
Groups:
- COPD-12 Sample With DMP Data: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with a follow-up of 12 months since index date and with available Data Monitoring Program (DMP) data (at least one entry during 3 months after index date).
Arm/Group | COPD-12 Sample | COPD-24 Sample | COPD-36 Sample | COPD-12 Sample With DMP Data
Number analyzed (Participants) | 14312 | 8804 | 3804 | 1434
Days | 123 [49 to 228] | 207 [74 to 417] | 287 [98 to 585] | 141 [60 to 245]

13. Secondary Outcome: Description of Direct Treatment Cost After Incident Diagnosis in COPD-12, COPD-24 and COPD-36 Samples
Description: Description of direct treatment cost in the first 12/24/36 months after incident diagnosis - yearly costs in incident chronic obstructive pulmonary disease (COPD) patients.
  LTOT: Long-Term Oxygen Therapy.
Time Frame: Up to 12, 24 and 36 months after index date for COPD-12, COPD-24 and COPD-36 sample respectively.
Population: Patients with newly diagnosed (incident) chronic obstructive pulmonary disease (COPD). Incident COPD-patients were reported by follow-up time (12, 24 and 36 months) and available Disease Management Program (DMP)-data. Arms are not mutually exclusive.
Measure: Number; unit: Euro per Person-year
Groups:
- COPD-12 Patients With Available DMP-data: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with a follow-up of 12 months since index date and with available Data Monitoring Program (DMP) data (at least one entry during 3 months after index date). (COPD DMP-12).
Arm/Group | COPD-12 Sample | COPD-24 Sample | COPD-36 Sample | COPD-12 Patients With Available DMP-data
Number analyzed (Participants) | 14213 | 8804 | 3804 | 1434
Euro per Person-year
  (Total) cost of outpatient visits (incl. costs for LTOT) | 1093.80 | 1059.52 | 1052.53 | 1179
  Total costs for GP visits | 456.77 | 446.63 | 444.03 | 429
  Total costs for pulmnologist visits | 72.52 | 67.30 | 61.67 | 185
  Total costs for other outpatient specialist visits | 564.51 | 545.59 | 546.82 | 565
  Inpatient cost (all-cause) | 10936.50 | 7013.81 | 5766.66 | 5508
  Total cost for hospitalizations with COPD-exacerbations | 398.86 | 228.28 | 165.79 | 414
  Total costs for hospitalizations with any COPD-diagnosis | 755.57 | 450.23 | 349.47 | 851
  Total costs for hospitalizations with any non-COPD-diagnosis | 10180.93 | 6563.58 | 5417.19 | 4657

14. Secondary Outcome: Prescription of Medication in COPD-12, COPD-24 and COPD-36 Samples
Description: Description of health-care resource use in the first 12/24/36 months after incident diagnosis - Prescription of medication.
  Top-5 prescription of non-COPD medication:
  Beta-blocking agents; Anti-thrombotic agents; Other analgesics & antipyretics; High-ceiling diuretics; Drugs for peptic ulcer or Gastroesophageal reflux disease (GERD).
  Other prescriptions:
  Antibiotics for systemic use (ATC J02AA); Antibiotics + corticosteroids (ATC D07C). Reported is number of yearly prescription.
Time Frame: Up to 12, 24 and 36 months after index date for COPD-12, COPD-24 and COPD-36 sample respectively.
Population: Patients with newly diagnosed (incident) chronic obstructive pulmonary disease (COPD). Incident COPD-patients were reported by follow-up time (12, 24 and 36 months). Arms are not mutually exclusive.
Measure: Mean (Standard Deviation); unit: Yearly prescription (of medication)
Groups:
- COPD-36 Sample: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2014 and march 2019, with a follow-up of 36 months since index date (COPD-36).
Arm/Group | COPD-12 Sample | COPD-24 Sample | COPD-36 Sample
Number analyzed (Participants) | 14213 | 8804 | 3804
Yearly prescription (of medication)
  Beta-blocking agents | 2.21 (2.49) | 2.16 (2.35) | 2.15 (2.29)
  Anti-thrombotic agents | 2.06 (3.00) | 1.87 (2.37) | 1.80 (2.16)
  Other analgesics & antipyretics | 1.07 (2.81) | 1.01 (2.43) | 0.93 (2.19)
  High-ceiling diuretics | 1.80 (2.55) | 1.67 (2.33) | 1.55 (2.21)
  Drugs for peptic ulcer or GERD | 1.59 (2.11) | 1.56 (1.94) | 1.58 (1.88)
  Antibiotics for systemic use | 0 (0) | 0.01 (0.02) | 0 (0)
  Antibiotics + corticosteroids (ATC D07C) | 0.03 (0.29) | 0.03 (0.24) | 0.03 (0.19)

15. Secondary Outcome: Number of Patients With Long Term Oxygen Therapy (LTOT) in COPD-12, COPD-24 and COPD-36 Samples
Description: Description of health-care resource use in the first 12/24/36 months after incident diagnosis - Number of Patients with Long Term Oxygen Therapy (LTOT).
Time Frame: Up to 12, 24 and 36 months after index date for COPD-12, COPD-24 and COPD-36 sample respectively.
Population: Patients with newly diagnosed (incident) chronic obstructive pulmonary disease (COPD). Incident COPD-patients were reported by follow-up time (12, 24 and 36 months).
Measure: Count of Participants; unit: Participants
Arm/Group | COPD-12 Sample | COPD-24 Sample | COPD-36 Sample
Number analyzed (Participants) | 14213 | 8804 | 3804
Participants | 2338 | 1696 | 741

16. Secondary Outcome: Time From Index Date Until Start of Long-term Oxygen Therapy (LTOT) - COPD-12, COPD-24 and COPD-36 Samples
Description: Time from index date until start of long-term oxygen therapy (LTOT) in days in the first 12/24/36 months after incident diagnosis.
Time Frame: Up to 12, 24 and 36 months after index date for COPD-12, COPD-24 and COPD-36 sample respectively.
Population: Patients with newly diagnosed (incident) chronic obstructive pulmonary disease (COPD). Incident COPD-patients were reported by follow-up time (12, 24 and 36 months) and available Disease Management Program (DMP) data. Only patients with any observed LTOT are included.
Measure: Mean (Standard Deviation); unit: Days
Groups:
- COPD-12 Sample With DMP Data: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with a follow-up of 12 months since index date and with available Disease Management Program (DMP) data (at least one entry during 3 months after index date). (COPD DMP-12).
- COPD-24 Sample With DMP Data: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with a follow-up of 24 months since index date and with available Disease Management Program (DMP) data (at least one entry during 3 months after index date). (COPD DMP-24).
- COPD-36 Sample With DMP Data: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with a follow-up of 36 months since index date and with available Disease Management Program (DMP) data (at least one entry during 3 months after index date). (COPD DMP-36).
Arm/Group | COPD-12 Sample | COPD-24 Sample | COPD-36 Sample | COPD-12 Sample With DMP Data | COPD-24 Sample With DMP Data | COPD-36 Sample With DMP Data
Number analyzed (Participants) | 2338 | 1696 | 741 | 269 | 223 | 93
Days | 68.9 (99.6) | 160.2 (214.4) | 88.6 (206.8) | 64.5 (100.4) | 159.1 (216.2) | 202.1 (294.6)

17. Secondary Outcome: Time From Index Date Until First Exacerbation - COPD-FULL, COPD-12, COPD-24 and COPD-36
Description: Time from index date until first exacerbation, in the first 12/24/36/48 months after incident diagnosis. Only severe exacerbations leading to an inpatient hospitalization after index date (documented as main diagnosis: ICD-10 J44.1) are considered.
Time Frame: Up to 12, 24, 36 and 48 months after index date for COPD-12, COPD-24, COPD-36 and COPD-FULL sample respectively.
Population: All patients with newly diagnosed (incident) chronic obstructive pulmonary disease. Incident COPD-patients were reported by follow-up time (12, 24, 36 and 48 months). Only patients with severe exacerbation leading to an inpatient hospitalization are included. Arms are not mutually exclusive.
Measure: Mean (Standard Error); unit: Months
Arm/Group | COPD-FULL Sample | COPD-12 Sample | COPD-24 Sample | COPD-36 Sample
Number analyzed (Participants) | 2102 | 1429 | 970 | 464
Months | 42.8 (0.1) | 42.9 (0.1) | 43.3 (0.2) | 43.5 (0.2)

18. Secondary Outcome: Average Number of Yearly Exacerbations During Follow-up - COPD-FULL, COPD-12, COPD-24 and COPD-36
Description: Average number of yearly exacerbations in the first 12/24/36 and 48 months after incident diagnosis.
Time Frame: Up to 12, 24, 36 and 48 months after index date for COPD-12, COPD-24, COPD-36 and COPD-FULL sample respectively.
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Exacerbations
Groups:
- COPD-FULL: Patients with incident chronic obstructive pulmonary disease (COPD) between April 2015 and March 2018 from German claims database were followed for up to 48 months. Patients were censored in case of death or loss to follow-up.
- COPD-12: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with a follow-up of 12 months since index date (COPD-12).
- COPD-24: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with a follow-up of 24 months since index date (COPD-24).
- COPD-36: Patients with chronic obstructive pulmonary disease (COPD) included in german claims database between april 2015 and march 2018, with a follow-up of 36 months since index date (COPD-36).
Arm/Group | COPD-FULL | COPD-12 | COPD-24 | COPD-36
Number analyzed (Participants) | 17464 | 14213 | 8804 | 3804
Exacerbations | 0.16 (0.57) | 0.14 (0.56) | 0.16 (0.64) | 0.18 (0.70)

19. Secondary Outcome: Average Medication Costs Per Year - COPD-12, COPD-24 and COPD-36
Description: Description of yearly costs in incident chronic obstructive pulmonary disease (COPD) patients.
  Cost of non-COPD-medication are based on the top-10 prescribed on non-COPD drug therapies.
Time Frame: Up to 12, 24 and 36 months after index date for COPD-12, COPD-24 and COPD-36 respectively.
Population: All patients with newly diagnosed (incident) chronic obstructive pulmonary disease. Incident COPD-patients are reported by follow-up time (12, 24 and 36 months). Arms are not mutually exclusive.
Measure: Mean (Standard Deviation); unit: Euro per Year (€/Y)
Arm/Group | COPD-12 Sample | COPD-24 Sample | COPD-36 Sample
Number analyzed (Participants) | 14213 | 8804 | 3804
Euro per Year (€/Y)
  Cost of COPD-medication (in total) | 317.46 (392.69) | 292.03 (367.37) | 273.50 (361.06)
  Cost of non-COPD-medication (in total) | 386.99 (713.16) | 355.92 (884.92) | 369.15 (2202.62)

ADVERSE EVENTS:
Time Frame: [All-cause Mortality]: Up to 48 months.
Description: [All-Cause Mortality]:Patients with newly diagnosed chronic obstructive pulmonary disease.
  As this is a non-interventional study with secondary use of data retrieved from a German claims database, safety monitoring and reporting on an individual case level is not applicable. Serious Adverse Events and Other Adverse Events are not collected in the database. "0" total Number of Participants at Risk means "Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed".
Arm/Group | COPD-FULL Sample
All-Cause Mortality (participants affected / at risk) | 5238/17464
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-16): https://cdn.clinicaltrials.gov/large-docs/23/NCT04097223/Prot_SAP_000.pdf